CLINICAL TRIAL: NCT01427803
Title: An Actual Use Trial In A Simulated OTC Environment of an Extended-Release Over-the-Counter NSAID
Brief Title: Actual Use Trial of Naproxen Sodium
Acronym: Kiefer AUT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15647
Record Dates: First submitted 2011-08-31; First posted 2011-09-02 (Estimated); Results first posted 2013-05-20 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2014-04

CONDITIONS: Pain
Keywords: Actual Use Trial
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Naproxen Sodium ER (BAYH6689)

INTERVENTIONS:
Drug: Naproxen Sodium ER (BAYH6689) — BAYH6689; oral tablet used as needed upon incidence of pain

SUMMARY:
An actual use trial to demonstrate that consumers will not exceed the labeled daily dose of Aleve 24 Hour at an unacceptable rate. Two aspects of consumer use will be evaluated: 1) the frequency at which consumers exceed the label-defined daily dose, thus putting themselves at clinical risk, and 2) the reasons for exceeding the labeled daily dose.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years of age
* Report taking OTC analgesics for pain on at least 5 days in the last month
* Report having had pain at least once in the last 3 months lasting longer than 12 hours or that they believe would have lasted longer than 12 hours if they had not treated it
* Able to read and understand English
* Provide written informed consent (subjects 12-17 years of age provide written assent and/or parent or legal guardian provide written consent)
* Provide contact information
* Purchase the investigational product

Exclusion Criteria:

* Have participated in a trial involving OTC analgesics in the last 6 months
* They or someone else in the household work for a market research company, an advertising agency, a public relations firm, a pharmaceutical company, as a healthcare professional, or as part of a health care practice (eliminated for reasons of confidentiality or increased awareness of drugs and their labels)
* Have a history of known allergies to NSAIDs (i.e., naproxen, ibuprofen, aspirin, etc.)
* Have a history of heart surgery in the last 60 days or plans for heart surgery in the next 60 days
* (Female subjects) are pregnant or breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 778 (Actual)
Dates: Start 2011-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (32):
- United States (32):
  - Hoover, Alabama
  - McCalla, Alabama
  - Pinson, Alabama
  - Mesa, Arizona
  - Anaheim, California
  - Oceanside, California
  - Yorba Linda, California
  - Overland Park, Kansas
  - Baltimore, Maryland
  - Andover, Minnesota
  - Elk River, Minnesota
  - Fridley, Minnesota
  - Northfield, Minnesota
  - Rosemount, Minnesota
  - Roseville, Minnesota
  - Kansas City, Missouri
  - Saint Joseph, Missouri
  - Savannah, Missouri
  - Albuquerque, New Mexico
  - Taos, New Mexico
  - Bountiful, Utah
  - Hurricane, Utah
  - Layton, Utah
  - Ogden, Utah
  - Salt Lake City, Utah
  - Syracuse, Utah
  - West Jordan, Utah
  - Montpelier, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Kenmore, Washington
  - Snohomish, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Patterns of Use Cohort: A subject was included in the Patterns of Use User Population if he/she completed the enrollment interview, purchased the investigational product, was randomized into the Patterns of Use Cohort, and provided e-diary data regarding their use.
- Reasons for Misuse Cohort: A subject was included in the Reasons for Misuse Interviewed Population if he/she completed the enrollment interview, purchased the investigational product, was randomized into the Reasons for Misuse Cohort, misused on one or more occasions (did not comply with the label directions [took more than one tablet per dose or a subsequent dose less than 22 hours later]), and completed the reasons for misuse questions.
Period: Overall Study
Arm/Group | Patterns of Use Cohort | Reasons for Misuse Cohort
Started | 526 | 252
Purchased Product | 525 (Only 516 participants used e-diary) | 252
Baseline Assessment | 516 | 130 (only interviewed participants were assessed)
Took Product | 508 (Those who took at least one dose of investigational product. Only 502 qualified for data analysis.) | 237 (Those who took at least one dose of investigational product as logged in e diary & 1 on Health Log.)
Completed | 463 | 226 (130 participants interviewed. Remaining subjects continued in trial to collect safety information.)
Not Completed | 63 | 26
Not completed — Lost to Follow-up | 32 | 26
Not completed — Withdrawal by Subject | 20 | 0
Not completed — Unable to complete full treatment period | 6 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 3 | 0
Not completed — did not take product | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patterns of Use User Population: A subject was included in the Patterns of Use User Population if he/she completed the enrollment interview, purchased the investigational product, was randomized into the Patterns of Use Cohort, and provided e-diary data regarding their use.
- Reasons for Misuse Interviewed Population: A subject was included in the Reasons for Misuse Interviewed Population if he/she completed the enrollment interview, purchased the investigational product, was randomized into the Reasons for Misuse Cohort, misused on one or more occasions (did not comply with the label directions [took more than one tablet per dose or a subsequent dose less than 22 hours later]), and completed the reasons for misuse questions.
- Total: Total of all reporting groups
Arm/Group | Patterns of Use User Population | Reasons for Misuse Interviewed Population | Total
Number analyzed (Participants) | 516 | 130 | 646
Age, Customized [Number; unit: Participants]
  12 to 17 Years | 3 | 0 | 3
  18 to 24 Years | 25 | 4 | 29
  25 to 34 Years | 63 | 13 | 76
  35 to 44 Years | 81 | 28 | 109
  45 to 54 Years | 142 | 30 | 172
  55 Years or Older | 202 | 55 | 257
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 295 | 68 | 363
  Male | 221 | 62 | 283

OUTCOME MEASURES:

1. Primary Outcome: Estimated Percentage of Misuse for Non-Therapeutic Reasons
Description: The primary objective of this trial was to determine the percentage of non-therapeutic misuse. Two aspects of consumer use of Aleve 24 Hour were examined: the frequency at which consumers exceeded the label-defined daily dose modified by those who did so for non-therapeutic reasons.
Time Frame: 28 days
Population: Participants in Patterns of Use cohort who took the product + Participants in Reason for Misuse cohort who completed interview
Measure: Number; unit: Percentage of Participants
Groups:
- Naproxen Sodium ER (BAYH6689): Subjects were allowed to purchase a maximum of two bottles of Naproxen Sodium ER during their participation in the trial. The package instructed subjects to take one tablet every 24 hours while symptoms lasted for no more than 10 consecutive days for pain and no more than three consecutive days for fever.
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 632
Percentage of Participants | 6.5

2. Secondary Outcome: Non-therapeutic Reasons for Misuse
Description: Those subjects in the Reasons for Misuse Cohort who did not state misuse due to need for additional pain relief were categorized to Non-therapeutic misuse.
Time Frame: 28 days
Population: Participants in Reason for Misuse cohort who misused the product due to non-therapeutic reasons were included in this analysis
Measure: Number; unit: Participants
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 130
Participants | 52

3. Secondary Outcome: Estimated Percentage of Misuse for Non-Therapeutic Reasons Using the First 10-Day Treatment Course
Description: This endpoint was an assessment of whether the rate of non-therapeutic misuse exceeded the pre-defined acceptable threshold for non-therapeutic misuse. The difference lay in the estimation of misuse in the Patterns of Use Cohort by using 10-day treatment courses rather than by "use day". A treatment course for each subject began on the first day they recorded taking one or more tablets which was followed by nine consecutive "evaluable days."
Time Frame: 28 days
Population: Participants in Patterns of Use cohort who took the product + Reasons for misuse interviewed population
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 632
Percentage of participants | 5

4. Secondary Outcome: Percentage of Participants Took >/= 2 Tablets/Use Day in Any 10 Use Days
Description: Percentage of participants took >/= 2 tablets/use day in any 10 use days thus exceeding the label directions during a treatment course.
Time Frame: 28 days
Population: Participants in Patterns of Use User Population who had at least 10 use days of the product
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 375
Percentage of participants | 14.9

5. Secondary Outcome: Percentage of Participants Who Took Product With Mean Daily Use >/= 2 Tablets /Use Day
Description: Percentage of participants who took product with mean daily use >/= 2 tablets /use day thus exceeding the label directions on any use day.
Time Frame: 28 days
Population: Participants in Patterns of Use User Population who had at least 10 use days of the product
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 375
Percentage of participants | 4.8

6. Secondary Outcome: Percentage of Participants With at Least One Dosing Occasion Where More Than One Tablet Was Taken
Description: Percentage of participants with at least one dosing occasion where more than one tablet was taken thus exceeding the label directions.
Time Frame: 28 days
Population: Participants in Patterns of Use cohort who took the product
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 502
Percentage of participants | 19.7

7. Secondary Outcome: Percentage of Dosing Occasions Where More Than One Tablet Was Taken
Description: Percentage of dosing occasions where more than one tablet was taken thus exceeding the label directions.
Time Frame: 28 days
Population: Participants in Patterns of Use cohort who took the product
Measure: Number; unit: Percentage of dosing occasions
Units Other Than Participants: Dosing occasions
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 502
Number analyzed (Dosing occasions) | 9895
Percentage of dosing occasions | 5.4

8. Secondary Outcome: Percentage of Participants Where a Dose Was Taken Less Than 22 Hours After the Most Recent Previous Dose
Description: Percentage of participants where a dose was taken less than 22 hours after the most recent previous dose thus exceeding the label directions. 22 hrs was chosen to allow for some imprecision in subjects' recollection.
Time Frame: 28 days
Population: Participants in Patterns of Use cohort who took the product
Measure: Number; unit: Percentage of participants
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 502
Percentage of participants | 72.5

9. Secondary Outcome: Percentage of Dosing Occasions Where a Dose Was Taken Less Than 22 Hours After the Most Recent Previous Dose
Description: Percentage of dosing occasions where a dose was taken less than 22 hours after the most recent previous dose. 22 hrs was chosen to allow for some imprecision in subjects' recollection
Time Frame: 28 days
Population: Participants in Patterns of Use cohort who took the product
Measure: Number; unit: Percentage of dosing occasions
Units Other Than Participants: Dosing occasions
Arm/Group | Naproxen Sodium ER (BAYH6689)
Number analyzed (Participants) | 502
Number analyzed (Dosing occasions) | 9895
Percentage of dosing occasions | 27.8

ADVERSE EVENTS:
Time Frame: 28 days
Description: AEs were collected at the Follow-up telephone interview after completion of the 28 day Use Phase or sooner if they discontinued from the study. The safety population consisted of all participants who took product. Safety data from the two cohorts were pooled in one group as both cohorts received the same treatment.
Arm/Group | Naproxen Sodium ER (BAYH6689)
Serious Adverse Events (participants affected / at risk) | 6/745
Other Adverse Events (participants affected / at risk) | 89/745
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium ER (BAYH6689) (N=745)
overdose (Injury, poisoning and procedural complications) | 1 (1)
cardiac failure congestive (Cardiac disorders) | 1 (1)
diarrhea haemorrhagic (Gastrointestinal disorders) | 1 (1)
viral infection (Infections and infestations) | 1 (1)
gallbladder disorder (Hepatobiliary disorders) | 1 (1)
hypersensitivity (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naproxen Sodium ER (BAYH6689) (N=745)
abdominal pain upper (Gastrointestinal disorders) | 14 (15)
constipation (Gastrointestinal disorders) | 12 (12)
diarrhoea (Gastrointestinal disorders) | 11 (11)
nasopharyngitis (Infections and infestations) | 20 (20)
headache (Nervous system disorders) | 14 (15)
sinusitis (Infections and infestations) | 10 (10)
back pain (Musculoskeletal and connective tissue disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days